CLINICAL TRIAL: NCT05623670
Title: Prospective Evaluation of Jugular Vein Thrombi After CPB Cervical Cannulation for Minimally Invasive Cardiac Surgery.
Brief Title: Prospective Evaluation of Jugular Vein Thrombi After CPB Cervical Cannulation
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, intensivist, Goethe University
Other Study IDs: VJI thrombi after CPB cervical
Record Dates: First submitted 2022-11-12; First posted 2022-11-21 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-01

CONDITIONS: Post-interventional VJI Thrombi After CPB

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients after minimally invasive cardiac surgery using a VJI cannula.
  Interventions: Procedure: minimally invasive cardiac surgery using a VJI cannula.

INTERVENTIONS:
Procedure: minimally invasive cardiac surgery using a VJI cannula. — Observation of postinterventional internal jugular vein thrombus after minimally invasive cardiac surgery using VJI cannulation to achieve complete CPB.

SUMMARY:
The primary objective of the study is to prospectively analyse the occurrence of post-interventional internal vena jugularis (VJI) thrombi after minimally invasive cardiac surgery using a VJI cannula to perform cardiopulmonary bypass (CPB). The study follows the question whether the performance of a jugular cannulation for the operation under CPB regularly causes wall thromboses despite continuous anticoagulation and a short length of stay of a few hours. The thromboses to be assessed for the study will be obtained by bedside (Doppler) sonography by experienced intensive care physicians in the cardiac surgery intensive care unit. A prospective analysis of all minimal invasive procedures performed with regard to thrombi in the VJI.

ELIGIBILITY:
Inclusion Criteria:

- Minimally invasive cardiac surgery carried out using complete cardiopulmonary bypass.

Exclusion Criteria:

* Postoperative support by veno-venous or veno-arterial extracorporeal membrane oxygenation.
* Complications of neck cannula placement or removal.
* Pre-existing occlusion of the vena jugularis interna
* Pre-existing thrombosis of the vena jugularis interna
* Pre-existing prothrombotic coagulation disorder
* Existing catheterisation of the vena jugularis interna within 14 days
* Pre-existing anatomical anomaly of the vena jugularis interna

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing minimally invasive cardiac surgery requiring full cardiopulmonary bypass at our centre during the observation period.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of post-interventional internal jugular vein thrombi | Detection of thrombi within 24 hours post-intervention
  Incidence of post-interventional internal jugular vein thrombi detectable by bedside (doppler) sonography by experienced intensivists in the cardiosurgical intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
Due to national legal restrictions, the publication of individual participant data is not possible without significant obstacles.